CLINICAL TRIAL: NCT03847350
Title: An Observational Study to Identify BEnefits After 24 Weeks of NEBILET®(Nebivolol) Administration For Essential hypertensIon Patients With Various Co-morbidities and Treatment Environments in KOREA.
Brief Title: Observational Study of Efficacy and Safety of Nebivolol in Korean Patients With Essential Hypertension
Acronym: BENEFIT
Status: Completed | Type: Observational
Sponsor: A.Menarini Asia-Pacific Holdings Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MAKR/15/Neb-Hyp/001
Record Dates: First submitted 2018-11-15; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is:

To evaluate the effects of NEBILET®(Nebivolol), used as monotherapy or in combination with other antihypertensive agents, in the control of BP and in the metabolic profile of patients with essential hypertension (with or without co-morbidities) after 12 weeks and 24 weeks.

DETAILED DESCRIPTION:
Nebivolol, the third-generation beta-blocker with vasodilatory effect, potentiates nitric oxide by activating the synthesis of nitric oxide of vascular endothelial cells and improves the function of vascular endothelial cells by reducing oxidation stress. The efficacy of NEBILET®(Nebivolol) has been demonstrated in randomized controlled trials not only as monotherapy but also as add-on therapy with angiotensin-converting-enzyme inhibitor, angiotensin II receptor blocker, diuretic and other anti-hypertensive agents in lowering the blood pressure.

Based on previous study results mentioned above, the present study aims to observe the effect of NEBILET®(Nebivolol) on controlling blood pressure and metabolic profile change in Korean patients with hypertension under routine clinical practice.

In addition, this study aims to identify additional benefits of NEBILET®(Nebivolol) administration in patients with essential hypertension under various treatment environments and existing co-morbidities in Korea, expected to provide detailed information about efficacy of blood pressure control, lipid and carbohydrate metabolism of NEBILET®(Nebivolol) administration in Korean patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient aged 19 and older
2. In patient diagnosed with essential hypertension,

   * Patients who can be first treated with NEBILET®(Nebivolol) to lower high blood pressure
   * In patients who are receiving other antihypertensive medications, those who can switch one of the antihypertensive agents to NEBILET®(Nebivolol) or use NEBILET®(Nebivolol) as an additional therapy (In case where one of other antihypertensive agents is switched to NEBILET®(Nebivolol), it is imperative that the dose of the previous medication should exhibit the same antihypertensive effect as NEBILET®(Nebivolol) 5 mg.)
3. Subjects who have signed the written informed consent form for their voluntary participation

Exclusion Criteria:

1. Patient with hypersensitivity to the NEBILET®(Nebivolol) substance
2. Patient with history of bronchospasm
3. Patient with history of bronchial asthma
4. Patient with metabolic acidosis
5. Patient with bradycardia(heart rate< 60 bpm)
6. Patient with second and third degree atrioventricular block
7. Patient with acute heart failure, cardiogenic shock, or episodes of heart failure decompensation requiring i.v. inotropic therapy)
8. Patient with uncontrolled severe heart failure
9. Patient with hypotension (Systolic Blood Pressure < 90mmHg)
10. Patient with severe peripheral circulatory disturbances
11. Patient with sick sinus syndrome including sino-atrial block
12. Patient with untreated pheochromocytoma
13. Patient with hepatic insufficiency
14. Patient with impaired liver function
15. Pregnant woman
16. Nursing mother
17. Patient with chronic heart failure who has severe renal insufficiency (serum creatinine ≥ 250 micro mol/L)
18. Patient with rare hereditary problems of galactose intolerance, the Lapp-lactase deficiency or glucose-galactose malabsorption
19. Patient who has participated in other clinical trial within the last 3 months

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female patient aged 19 and older
Study Population: Male and female patients with essential hypertension
Sampling Method: Probability Sample
Enrollment: 3250 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Mean change of the Systolic Blood Pressure and Diastolic Blood Pressure | 24 weeks
  Mean change of the Systolic Blood Pressure and Diastolic Blood Pressure after 12 weeks(±2 weeks) and 24 weeks (±2 weeks) compared to Baseline

SECONDARY OUTCOMES:
Controlled patient rate in targeted Systolic Blood Pressure and Diastolic Blood Pressure range | 24 weeks
  Controlled patient rate in targeted Systolic Blood Pressure and Diastolic Blood Pressure range after 12 weeks (±2 weeks) and 24 weeks (±2 weeks) compared to Baseline
Change of glucose (HbA1c, fasting blood sugar), Na, K, total cholesterol, triglyceride, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol | 24 weeks
  Change of glucose (HbA1c, fasting blood sugar), Na, K, total cholesterol, triglyceride, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol at 12 weeks (±2 weeks) and 24 weeks (±2 weeks) compared to Baseline
Changes in Heart Rate and Heart Rate Variability after treatment with NEBILET® (Nebivolol) versus baseline values in patients receiving the concomitant antihypertensive therapies. | 24 weeks
  Changes in Heart Rate and Heart Rate Variability at 12 weeks (±2 weeks) and 24 weeks (±2 weeks) after treatment with NEBILET® (Nebivolol) versus baseline values in patients receiving the concomitant antihypertensive therapies.
Mean change of the Systolic Blood Pressure and Diastolic Blood Pressure compared to baseline depending on the treatment status and type of anti-hypertensive concomitant medication | 24 weeks
  Mean change of the Systolic Blood Pressure and Diastolic Blood Pressure after 12 weeks and 24 weeks compared to baseline depending on the treatment status and type of anti-hypertensive concomitant medication

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Hyeok Kim, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munzel T, Gori T. Nebivolol: the somewhat-different beta-adrenergic receptor blocker. J Am Coll Cardiol. 2009 Oct 13;54(16):1491-9. doi: 10.1016/j.jacc.2009.05.066. PMID 19815121
- [Background] Neutel JM, Smith DH, Gradman AH. Adding nebivolol to ongoing antihypertensive therapy improves blood pressure and response rates in patients with uncontrolled stage I-II hypertension. J Hum Hypertens. 2010 Jan;24(1):64-73. doi: 10.1038/jhh.2009.33. PMID 19404314
- [Background] Badar VA, Hiware SK, Shrivastava MP, Thawani VR, Hardas MM. Comparison of nebivolol and atenolol on blood pressure, blood sugar, and lipid profile in patients of essential hypertension. Indian J Pharmacol. 2011 Jul;43(4):437-40. doi: 10.4103/0253-7613.83117. PMID 21845001
- [Background] Predel HG, Mainka W, Schillings W, Knigge H, Montiel J, Fallois J, Agrawal R, Schramm T, Graf C, Giannetti BM, Bjarnason-Wehrens B, Prinz U, Rost RE. Integrated effects of the vasodilating beta-blocker nebivolol on exercise performance, energy metabolism, cardiovascular and neurohormonal parameters in physically active patients with arterial hypertension. J Hum Hypertens. 2001 Oct;15(10):715-21. doi: 10.1038/sj.jhh.1001257. PMID 11607802
- [Background] Van Bortel LM. Efficacy, tolerability and safety of nebivolol in patients with hypertension and diabetes: a post-marketing surveillance study. Eur Rev Med Pharmacol Sci. 2010 Sep;14(9):749-58. PMID 21061833
- [Background] Okamoto LE, Gamboa A, Shibao CA, Arnold AC, Choi L, Black BK, Raj SR, Robertson D, Biaggioni I. Nebivolol, but not metoprolol, lowers blood pressure in nitric oxide-sensitive human hypertension. Hypertension. 2014 Dec;64(6):1241-7. doi: 10.1161/HYPERTENSIONAHA.114.04116. Epub 2014 Sep 29. PMID 25267802
- [Background] Neutel JM, Giles TD, Punzi H, Weiss RJ, Li H, Finck A. Long-term safety of nebivolol and valsartan combination therapy in patients with hypertension: an open-label, single-arm, multicenter study. J Am Soc Hypertens. 2014 Dec;8(12):915-20. doi: 10.1016/j.jash.2014.09.017. Epub 2014 Sep 28. PMID 25492835
- [Background] Punzi H, Lewin A, Lukic T, Goodin T, Wei Chen. Efficacy and safety of nebivolol in Hispanics with stage I-II hypertension: a randomized placebo-controlled trial. Ther Adv Cardiovasc Dis. 2010 Dec;4(6):349-57. doi: 10.1177/1753944710387629. PMID 21088095
- [Derived] Shin J, Cha DH, Bae WH, Jung IH, Hong SP, Kim SH, Do JY, Hwang WM, Koh YY, Mancia G, Manolis AJ, Lee M. Posttreatment pulse rate reduction and not baseline pulse rate as an indicator of blood pressure response to nebivolol: a subanalysis from the real-world BENEFIT-KOREA study. Clin Hypertens. 2025 Mar 1;31:e8. doi: 10.5646/ch.2025.31.e8. eCollection 2025. PMID 40083595
- [Derived] Cho KI, Jeon DW, Ahn HS, Jin DK, Lee HS, Lee JY, Lim HS, Manolis AJ, Rha SW, Park SW. Efficacy and safety of nebivolol in Korean patients with hypertension by age and sex: a subanalysis from the BENEFIT-KOREA study. Clin Hypertens. 2021 Mar 15;27(1):9. doi: 10.1186/s40885-021-00165-3. PMID 33722290
- [Derived] Shin J, Choi YJ, Hong GR, Jeon DW, Kim DH, Koh YY, Mancia G, Manolis AJ, Yoon HJ, Park SW. Real-world efficacy and safety of nebivolol in Korean patients with hypertension from the BENEFIT KOREA study. J Hypertens. 2020 Mar;38(3):527-535. doi: 10.1097/HJH.0000000000002296. PMID 31693535